CLINICAL TRIAL: NCT05363501
Title: Single Dose, Crossover, Pharmacokinetic Evaluation of a New Naloxone Nasal Swab, Naloxone Nasal Spray, and Intramuscular Naloxone Injection in Healthy Volunteers
Brief Title: Pharmacokinetic Evaluation of a New Naloxone Nasal Swab, Naloxone Nasal Spray, and Intramuscular Naloxone Injection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pocket Naloxone Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PNC-20-001
Record Dates: First submitted 2022-04-04; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-12

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Naloxone IM Injection (Active Comparator): Single 0.4 mg IM naloxone injection will be administered (1 mL of 0.4 mg/mL injection, into the gluteus maximus muscle using a 23-gauge needle).
  Interventions: Drug: IM Naloxone Injection
- Intranasal Naloxone Spray (Active Comparator): Single 4 mg intranasal naloxone spray will be administered in one nostril (0.1 mL of 4 mg/0.1 mL spray, based on the prescribing information and approved Instructions for Use).
  Interventions: Drug: Naloxone Nasal Spray
- Single 8 mg naloxone nasal swab-Swirl method (Experimental): Single 8 mg naloxone nasal swab administered as one swab in one nostril, swirled 3 times around the inside of the nasal mucosa.
  Interventions: Drug: Naloxone Nasal Swab
- Single 4 mg naloxone nasal swab-Swirl method (Experimental): Single 4 mg naloxone nasal swab administered as one swab in one nostril, swirled 3 times around the inside of the nasal mucosa.
  Interventions: Drug: Naloxone Nasal Swab
- Single 12 mg naloxone nasal swab-Swirl method (Experimental): Single 12 mg naloxone nasal swab administered as one swab in one nostril, swirled 3 times around the inside of the nasal mucosa.
  Interventions: Drug: Naloxone Nasal Swab
- Single 12 mg naloxone nasal swab-Squeeze method (Experimental): Single 12 mg naloxone nasal swab administered into the nasal cavity - administered in one nostril and using two fingers to squeeze outside of both nostrils.
  Interventions: Drug: Naloxone Nasal Swab
- Single 12 mg naloxone nasal swab in each nostril-Squeeze method (Experimental): Two 12 mg naloxone nasal swabs in both nostrils- administered one per nostril and using two fingers to squeeze outside of both nostrils (two doses given sequentially)
  Interventions: Drug: Naloxone Nasal Swab
- Single 8 mg naloxone nasal swab in each nostril-Squeeze method (Experimental): Two 8 mg naloxone nasal swab in both nostrils - administered one per nostril and using two fingers to squeeze outside of both nostrils (two doses given sequentially)
  Interventions: Drug: Naloxone Nasal Swab
- Single 12.5 mg naloxone nasal swab-Squeeze method (Experimental): Single target naloxone nasal swab dose identified in Phase 1(12.5 mg) administered as one swab in one nostril, using the insert into nostril and squeeze method of administration
  Interventions: Drug: Naloxone Nasal Swab
- Single 12.5 mg naloxone nasal swab in each nostril-Squeeze method (Experimental): Single target naloxone nasal swab dose identified in Phase 1 (12.5 mg) using the insert into each nostril and squeeze method of administration (two doses given in total).
  Interventions: Drug: Naloxone Nasal Swab

INTERVENTIONS:
Drug: IM Naloxone Injection — Single 0.4 mg IM naloxone injection will be administered (1 mL of 0.4 mg/mL injection, into the gluteus maximus muscle using a 23-gauge needle).
  Arms: Naloxone IM Injection
Drug: Naloxone Nasal Spray — Single 4 mg intranasal naloxone spray will be administered in one nostril (0.1 mL of 4 mg/0.1 mL spray, based on the prescribing information and approved Instructions for Use).
  Arms: Intranasal Naloxone Spray
Drug: Naloxone Nasal Swab — 4 mg naloxone nasal swab administered in nostril
  Arms: Single 4 mg naloxone nasal swab-Swirl method
Drug: Naloxone Nasal Swab — 8 mg naloxone nasal swab administered in nostril
  Arms: Single 8 mg naloxone nasal swab in each nostril-Squeeze method; Single 8 mg naloxone nasal swab-Swirl method
Drug: Naloxone Nasal Swab — 12 mg naloxone nasal swab administered in nostril
  Arms: Single 12 mg naloxone nasal swab in each nostril-Squeeze method; Single 12 mg naloxone nasal swab-Squeeze method; Single 12 mg naloxone nasal swab-Swirl method
Drug: Naloxone Nasal Swab — 12.5 mg naloxone nasal swab administered in nostril
  Arms: Single 12.5 mg naloxone nasal swab in each nostril-Squeeze method; Single 12.5 mg naloxone nasal swab-Squeeze method

SUMMARY:
The study consists of two Phases with the first phase (Pilot Phase) divided into two sub phases.

In each study phase, subjects will be admitted to the clinical unit from 10 hours prior to the first drug administration on Day -1 until approximately 12 hours following the last study drug administration. Screening of alcohol and drugs of abuse will be performed before the first study drug administration. For female subjects, a pregnancy test will be performed before the first drug administration. Clinical nasal irritation rating and the Brief Smell Identification Test will be performed at screening.

DETAILED DESCRIPTION:
The study consists of two Phases with the first phase (Pilot Phase) divided into two sub phases.

In each study phase, subjects will be admitted to the clinical unit from 10 hours prior to the first drug administration on Day -1 until approximately 12 hours following the last study drug administration. Screening of alcohol and drugs of abuse will be performed before the first study drug administration. For female subjects, a pregnancy test will be performed before the first drug administration. Clinical nasal irritation rating and the Brief Smell Identification Test will be performed at screening.

Phases 1A and , 1B, and 1C (Pilot Phase) The first sub-phase, Phase 1A, will be an inpatient, 5-period, 5-treatment, crossover study involving 10 healthy subjects.

In Phase 1A of the study, qualified subjects will receive one of the following treatment in the morning, after a 10 hour overnight fast:

* Treatment-1: Single 0.4 mg IM naloxone injection will be administered (1 mL of 0.4 mg/mL injection, into the gluteus maximus muscle using a 23-gauge needle).
* Treatment-2: Single 4 mg intranasal naloxone spray will be administered in one nostril (0.1 mL of 4 mg/0.1 mL spray, based on the prescribing information and approved Instructions for Use).
* Treatment-3: Single 8 mg naloxone nasal swab administered as one swab in one nostril, swirled 3 times around the inside of the nasal mucosa.
* Treatment-4: Single 4 mg naloxone nasal swab administered as one swab in one nostril, swirled 3 times around the inside of the nasal mucosa.
* Treatment-5: Single 12 mg naloxone nasal swab administered as one swab in one nostril, swirled 3 times around the inside of the nasal mucosa.

Based on preliminary results from Phase 1A, additional administration technique and higher dose will be tested. The second sub-phase, Phase 1B, will be a separate inpatient crossover study involving 10 healthy subjects which will start after completion of Phase 1A. Every attempt will be made to include the same subjects from Phase 1A in Phase 1B.

In Phase 1B of the study, qualified subjects will receive one of the following treatments in the morning, after a 10 hour overnight fast:

* Treatment-1: Single 12 mg naloxone nasal swab administered into the nasal cavity - administered in one nostril and using two fingers to squeeze outside of both nostrils.
* Treatment-2: Two 12 mg naloxone nasal swabs in both nostrils- administered one per nostril and using two fingers to squeeze outside of both nostrils (two doses given sequentially)
* Treatment-3: Two 8 mg naloxone nasal swab in both nostrils - administered one per nostril and using two fingers to squeeze outside of both nostrils (two doses given sequentially) For all intranasal treatments (nasal spray and nasal swab), participants will be instructed to not breathe through the nose during treatment administration. The same nostril will be used throughout the study for all nasal treatments requiring one nostril only administration. If a Coronavirus Disease 2019 (COVID-19) test is performed prior to administration, the opposite nostril will be used for administration for treatments requiring one nostril administration.

The order in which subjects receive their treatment will not be randomized. During Phase 1A, subjects will receive Treatment-1 in period 1, Treatment-2 in period 2, Treatment-3 in period 3, Treatment-4 in period 4, and Treatment-5 in period 5. In Phase 1B, subjects will receive Treatment-1 in period 1, Treatment-2 in period 2, and Treatment-3 in period 3. There will be a 4 day wash out window between treatment periods. At the end of Phase 1A and Phase 1B, a dose will be selected as the proposed target dose for the Phase 2 to confirm the PK profiles.

Phase 2 (Confirmatory Phase)

Phase 2 of the study will be an inpatient, randomized, laboratory-blinded, balanced, 4-way (4 treatments) crossover study with 4 sequences (Williams design). Below are the 4 treatments to be utilized:

* Treatment-1: Single target naloxone nasal swab dose identified in Phase 1 (12.5 mg) administered as one swab in one nostril, using the insert into nostril and squeeze method of administration.
* Treatment-2: Single target naloxone nasal swab dose identified in Phase 1 (12.5 mg) using the insert into each nostril and squeeze method of administration (two doses given in total).
* Treatment-3: Single 0.4 mg IM naloxone injection will be administered (1 mL of 0.4 mg/mL injection, into the gluteus maximus muscle using a 23-gauge needle).
* Treatment-4: Single 4 mg intranasal naloxone spray will be administered in one nostril (0.1 mL of 4 mg/0.1 mL spray, based on the prescribing information and approved Instructions for Use) For all intranasal treatments (nasal spray and nasal swab), participants will be instructed to not breathe through the nose during treatment administration. The same nostril will be used throughout the study for all nasal treatments except Treatment-2 where the swab administered in both nostrils. If a COVID-19 test is performed prior to administration, the opposite nostril will be used for administration of all single swab or spray doses.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy adult male or female
4. If female, meets 1 of the following criteria:

   1. Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include:

      * Abstinence from heterosexual intercourse from the first study drug administration through to at least 30 days after the last dose of the study drug
      * 1 of the following highly-effective contraceptive methods, used from at least 28 days prior to the first study drug administration through to at least 30 days after the last dose of the study drug: Systemic contraceptives (combined birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch) Intrauterine device (with or without hormones) Male partner vasectomized at least 6 months prior to the first study drug administration
      * The following effective contraceptive method, used from the first study drug administration through to at least 30 days after the last dose of the study drug:

      Male condom with diaphragm/cervical cap plus spermicide Or
   2. Male partner has had a vasectomy less than 6 months prior to dosing, and the female subject agrees to use an additional acceptable contraceptive method from the first study drug administration through to at least 30 days after the last dose of the study drug Or
   3. Is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study drug administration)
5. Aged at least 18 years but not older than 55 years
6. Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
7. Non- or ex-smoker (An ex smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
8. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs), ECG, and/or nasal cavity examination, as determined by an investigator

Exclusion Criteria:

1. Female who is lactating at screening
2. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. Seated blood pressure higher than 140/90 mmHg at screening or prior to the first study drug administration
4. History of significant hypersensitivity to naloxone or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
5. Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
6. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
7. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment
8. Any intranasal conditions including nostril piercing, abnormal nasal anatomy, nasal symptoms (i.e., blocked and/or runny nose, nasal polyps, etc.), or having a product sprayed into the nasal cavity prior to drug administration
9. Current or recent upper respiratory tract infection (within 28 days before the first study drug administration)
10. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
11. Any clinically significant illness in the 28 days prior to the first study drug administration
12. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the participant as healthy
13. Any history of tuberculosis
14. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
15. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus antibody tests
16. Any other clinically significant abnormalities at screening that would, in the opinion of an investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
17. Inclusion in a previous group for this clinical study (for Phase 2 only)
18. Intake of naloxone in the 28 days prior to the first study drug administration
19. Intake of an Investigational Product (IP) in the 28 days prior to the first study drug administration
20. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
21. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — For Phase 2, at least 20% of each gender are included in the trial.
Enrollment: 76 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Various Naloxone Administrations (Maximum plasma concentration (Cmax))-Phase 1 | 17 days
  To determine the pharmacokinetics (PK) of various naloxone intranasal swab doses (4, 8, and 12 mg) compared to intramuscular (IM) naloxone injection (0.4 mg dose) and naloxone nasal spray (4 mg dose) in healthy subjects. Maximum plasma concentration (Cmax) will be measured.
Pharmacokinetics of Various Naloxone Administrations (Area Under the Curve (AUC))-Phase 1 | 17 days
  To determine the pharmacokinetics (PK) of various naloxone intranasal swab doses (4, 8, and 12 mg) compared to intramuscular (IM) naloxone injection (0.4 mg dose) and naloxone nasal spray (4 mg dose) in healthy subjects. Area Under the Curve (AUC)will be measured.
Pharmacokinetics of Various Naloxone Administrations (Partial Area Under the Curve (AUC))-Phase 1 | 17 days
  To determine the pharmacokinetics (PK) of various naloxone intranasal swab doses (4, 8, and 12 mg) compared to intramuscular (IM) naloxone injection (0.4 mg dose) and naloxone nasal spray (4 mg dose) in healthy subjects. Partial Area Under the Curve (AUC) will be measured.
Dose Selection (Maximum plasma concentration (Cmax))-Phase 1 | 17 days
  To identify an appropriate target intranasal swab dose using comparative PK parameters with IM naloxone injection (0.4 mg) and naloxone nasal spray (4 mg dose) in healthy subjects.
  Maximum plasma concentration (Cmax) will be measured.
Dose Selection (Area Under the Curve (AUC))-Phase 1 | 17 days
  To identify an appropriate target intranasal swab dose using comparative PK parameters with IM naloxone injection (0.4 mg) and naloxone nasal spray (4 mg dose) in healthy subjects. Area Under the Curve (AUC) will be measured.
Dose Selection (Partial Area Under the Curve (AUC))-Phase 1 | 17 days
  To identify an appropriate target intranasal swab dose using comparative PK parameters with IM naloxone injection (0.4 mg) and naloxone nasal spray (4 mg dose) in healthy subjects. Partial Area Under the Curve (AUC) will be measured.
Bioavailability (Maximum plasma concentration (Cmax))-Phase 2 | 13 days
  To evaluate and compare the bioavailability of the identified nasal naloxone swab target dose from the Phase 1 (12.5 mg) and IM naloxone injection (0.4 mg). Maximum plasma concentration (Cmax) will be measured.
Bioavailability (Area Under the Curve (AUC))-Phase 2 | 13 days
  To evaluate and compare the bioavailability of the identified nasal naloxone swab target dose from the Phase 1 (12.5 mg) and IM naloxone injection (0.4 mg). Area Under the Curve (AUC) will be measured.
Bioavailability (Partial Area Under the Curve (AUC))-Phase 2 | 13 days
  To evaluate and compare the bioavailability of the identified nasal naloxone swab target dose from the Phase 1 (12.5 mg) and IM naloxone injection (0.4 mg). Partial Area Under the Curve (AUC) will be measured.

SECONDARY OUTCOMES:
Absorption Levels-Phase 1 and 2 | 17 days
  To compare the absorption levels of intranasal naloxone swab at early time points post -delivery (within the first 15 minutes) with IM naloxone injection (0.4 mg) and naloxone nasal spray (4 mg dose) in healthy subjects.
Safety of Naloxone Swab- (Treatment emergent adverse events (TEAEs))-Phase 1 and 2 | 17 days
  To determine the safety and tolerability of intranasal naloxone swab doses (4, 8, 12 and 12.5 mg), particularly with respect to nasal irritation (erythema, edema, and erosion) and olfactory nerve abnormalities in healthy subjects. will be included in the adverse event summaries.
Absorption Levels-Phase 2 | 13 days
  To compare the absorption levels of the nasal swab at early time points post-delivery (within the first 15 minutes) with IM naloxone injection (0.4 mg) and naloxone nasal spray (4 mg dose) in healthy subjects.
Dose Proportionality-Phase 2 | 13 days
  To evaluate the dose proportionality of naloxone nasal swab target dose (12.5 mg).

CONTACTS AND LOCATIONS:
Overall Officials: Sonnie Kim, Study Director — Pocket Naloxone Corp
Locations (1):
- Altasciences, Québec, Quebec, Canada